CLINICAL TRIAL: NCT03638375
Title: Adoptive TIL Therapy With Low-dose IFN-alpha Plus Anti-PD1 in Metastatic Melanoma
Brief Title: TIL and Anti-PD1 in Metastatic Melanoma
Acronym: ACTME
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Leiden University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, HW Kapiteijn, Principal Investigator, Leiden University Medical Center
Organization: Leiden University Medical Center (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NL64805.000.18
Record Dates: First submitted 2018-07-05; First posted 2018-08-20 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Toxicity, Drug; Adverse Drug Event; Effects of Immunotherapy
Keywords: Metastatic melanoma; anti-PD1; TIL; interferon-alpha; adoptive cell therapy; nivolumab
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Melanoma | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: The ACTME trial consists of both a phase I part to determine safety and feasibility and a phase II part to evaluate first clinical activity of IFN-alpha, nivolumab and TIL. The treatment with IFN-alpha will be added after the combination of TIL and nivolumab has proven to be safe.
  Phase 1, Cohort 1: Adding TIL therapy to anti-PD1 immunotherapy. Phase 1, Cohort 2: Adding IFN-alpha to the treatment with TIL and anti-PD1 immunotherapy.
  Phase 2: Patients will be treated with TIL, IFN-alpha and anti-PD1 according to the same schedule as used in phase 1 cohort 2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment with nivolumab plus TIL (Experimental): In the first cohort the subcutaneous IFN-alpha injections will be omitted and the combination of nivolumab and TIL is given.
  * Nivolumab is given 3mg/kg i.v. once every two weeks and starts 4 weeks before the first TIL infusion
  * TILs are given at a dose ranging between 2.5-7.5x10^8 T cells i.v. once every three weeks, three times per cycle.
  Interventions: Drug: Nivolumab & Tumor Infiltrating Lymphocytes with/without Interferon-Alpha
- Treatment with Nivolumab plus TIL and IFN-alpha (Experimental): In the second cohort of the first phase and the second phase of the trial patients will be treated with subcutaneous IFN-alpha injections in combination with TIL and nivolumab.
  * IFN-alpha is given at a fixed dose of 3 million IU s.c. every day, for 11 weeks, starting one week before the first TIL infusion
  * Nivolumab is given 3mg/kg i.v. once every two weeks and starts 4 weeks before the first TIL infusion
  * TILs are given at a dose ranging between 2.5-7.5x10^8 T cells i.v. once every three weeks, three times per cycle.
  Interventions: Drug: Nivolumab & Tumor Infiltrating Lymphocytes with/without Interferon-Alpha

INTERVENTIONS:
Drug: Nivolumab & Tumor Infiltrating Lymphocytes with/without Interferon-Alpha — During 15 weeks patients will be treated with nivolumab (3mg/kg i.v.) once every two weeks. Four weeks after starting nivolumab, patients will receive their first TIL infusion (2.5-7.5x10^8 T cells i.v.) once every three weeks for three infusions.
  In the second group treatment with IFN-alpha (3 million IU s.c.) daily will be added one week before the first TIL infusion and will be continued for 11 weeks.

SUMMARY:
The ACTME study is an investigator initiated, single center phase I/II clinical trial for patients with progressive unresectable stage III or stage IV melanoma. The trial consists of both a phase I part to determine safety and feasibility and a phase II part to evaluate first clinical activity of IFN-alpha, nivolumab and TIL. The treatment with IFN-alpha will be added after the combination of TIL and nivolumab has proven to be safe.

DETAILED DESCRIPTION:
The ACTME is an investigator initiated, single center phase I/II clinical trial for patients with progressive unresectable stage III or stage IV melanoma.

Patients are conditioned by low-dose IFN-alpha and treated with ACT and PD-1 antibodies. With this approach the investigators hope to solve 4 of the most important aspects curtailing the efficacy of current immunotherapies in metastatic melanoma:

1. the lack of sufficient numbers of activated tumor-reactive T cells in patients by providing ACT; and
2. the inhibition of T-cell effector function through PD-1 signalling by administration of nivolumab; as well as
3. the toxicity of high-dose IL-2, and
4. long term hospitalization of patients due to the conditioning-regimen used in most ACT protocols by replacing it with low-dose IFN-alpha treatment.

The trial consists of both a phase I part to determine safety and feasibility and a phase II part to evaluate first clinical activity of IFN-alpha, nivolumab and TIL.

The treatment with IFN-alpha will be added after the combination of TIL and nivolumab has proven to be safe in the first cohort of the phase I part of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Histologically or cytologically proven metastatic skin melanoma
3. Melanoma must be at one of the following AJCC 2009 stages:

   * Unresectable (or residual) regional metastatic melanoma, i.e. in terms of AJCC 2009 classification unresectable stage III melanoma, or
   * Stage IV melanoma, i.e. distant metastatic disease (any T, any N, M1a, M1b or M1c), and normal LDH
   * Patients have failed on standard treatment options
4. Patients with brain metastases have to be neurologically stable for at least 2 months and should not use dexamethasone
5. Presence of measurable progressive disease according to RECIST version 1.1
6. Expected survival of at least 3 months
7. WHO performance status ≤1
8. Within the last 2 weeks prior to study day 1, vital laboratory parameters should be within normal range, except for the following laboratory parameters, which should be within the ranges specified:

   Lab Parameter Range Hemoglobin ≥ 6,0 mmol/l Granulocytes ≥ 1,500/µl Lymphocytes ≥ 700/µl Platelets ≥ 100,000/µl Creatinine clearance ≥ 60 min/ml Serum bilirubin ≤ 40 µmol/l ASAT and ALAT ≤ 5 x the normal upper limit LDH ≤ 2 x the normal upper limit
9. Viral tests must be performed at least 30 days before surgery:

   * Negative for HIV type 1/2, HTLV and TPHA
   * No HBV (hepatitis B virus) antigen or antibodies against HBc in the serum
   * No antibodies against HCV (hepatitis C virus) in the serum
10. Able and willing to give valid written informed consent.
11. Progressive disease on prior treatment with f.e. BRAF-inhibitors, MEK-inhibitors or immunotherapy, including anti-PD1 treatment. Systemic therapy must have been discontinued for at least four weeks before start of study treatment.

Exclusion Criteria:

1. Patients with brain metastases who are neurologically unstable and/or use dexamethasone
2. Clinically significant heart disease (NYHA Class III or IV)
3. Other serious acute or chronic illnesses, e.g. active infections requiring antibiotics, bleeding disorders, or other conditions requiring concurrent medications not allowed during this study
4. Active immunodeficiency disease, autoimmune disease requiring immune suppressive drugs or autoimmune adverse events following treatment with checkpoint inhibitors. Vitiligo is not an exclusion criterion
5. Subjects with a condition requiring systemic chronic steroid therapy (≥ 10mg/day prednisone or equivalent) or any immunosuppressive therapy within 14 days prior to planned date for first dose of study treatment. Topical, inhaled, nasal and ophthalmic steroids, and adrenal replacement therapy are allowed.
6. Other malignancy within 2 years prior to entry into the study, except for treated non-melanoma skin cancer and in situ cervical carcinoma
7. Mental impairment that may compromise the ability to give informed consent and comply with the requirements of the study
8. Any serious or uncontrolled medical disorder or active infection that, in the opinion of the investigator, may increase the associated with the participation, study drug administration, or would impair the ability of the patient to receive protocol therapy
9. Lack of availability for follow-up assessments
10. Pregnancy or breastfeeding
11. Known allergy to penicillin or streptomycin (used during the culturing of T cells)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2018-07-31 (Actual); Primary Completion 2025-11-29 (Estimated); Study Completion 2025-11-29 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related serious adverse events as assessed by CTCAE 4.0 criteria | 14 weeks after start of treatment
  To evaluate the safety and toxicity of ACT with nivolumab, followed by evaluating the safety and toxicity of IFN-alpha, and nivolumab plus ACT according to the common terminology criteria of adverse events (CTCAE) 4.0 criteria. Treatment related adverse events grade 3 or less and SAE related to treatment that do not result in treatment termination are considered acceptable for continuation of the study.
  * Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  * Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL
  * Grade 3: Severe or medically significant but not immediately life-threatening hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL
  * Grade 4: Life-threatening consequences; urgent intervention indicated
  * Grade 5: Death related to AE

SECONDARY OUTCOMES:
Evaluation of disease control rate according to RECIST 1.1 criteria | 14 weeks after first nivolumab infusion
  Disease control is defined by complete response, partial response or stable according to RECIST 1.1 versus no clinical benefit defined as progressive disease.
  Complete response: Disappearance of all target and nontarget lesions, nodes must regress to <10mm short axis, no new lesions, confirmation required Partial response: ≥30% decrease in tumor burden compared with baseline, confirmation required Progressive disease: ≥20% + 5 mm absolute increase in tumor burden compared with nadir, appearance of new lesions or progression of nontarget lesions Stable disease: neither partial response nor progressive disease
Evaluation of disease control rate according to immune RECIST response criteria | 14 weeks after first nivolumab infusion
  Disease control is defined by complete response, partial response or stable according to the iRECIST versus no clinical benefit defined as progressive disease.
  Complete response: Disappearance of all lesions Partial response: ≥30% decrease in tumor burden compared with baseline. Progressive disease: ≥20% + 5 mm absolute increase in tumor burden compared with nadir Stable disease: neither progressive disease nor partial response
To study the potential working mechanisms of the different treatment compounds. Therefore, blood will be drawn to analyse changes in circulating immune cells and their function during treatment. | Within 5 years after first inclusion
  The investigators will analyse the patients their tumor material, blood, serum and the TILs used for infusion
To establish a possible prognostic biomarker profile in patients tumor material, blood, serum and TILs used for infusion | Within 5 years after first inclusion
  The investigators will analyse the patients their tumor material, blood, serum and the TILs used for infusion to look at changes in the number and phenotype of circulating immune cells, the cytokines that are produced by these cells and serum/plasma markers of persistence.
To characterize the infusion product | Within 5 years after first inclusion
  The expression of co-inhibitory molecules on T cells and regulatory T cells will be measured by flow cytometry. Furthermore, the investigators will assess the fraction of tumor-specific TIL, their cytolytic capacity as well as to analyse their persistence in the circulation. The supernatants of T cell are used for cytokine analysis assays.
To analyse potential correlations between the clinical response and hypothesis related immune parameters | Within 5 years after first inclusion
To analyse the overall survival following treatment | Within 5 years after first inclusion
  The overall survival of all patients entering the study will be monitored

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Kapiteijn, Dr., Principal Investigator — LUMC
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van der Kooij MK, Verdegaal EME, Visser M, de Bruin L, van der Minne CE, Meij PM, Roozen ICFM, Jonker MA, van den Bosch S, Liefers GJ, Speetjens FM, van der Burg SH, Kapiteijn E. Phase I/II study protocol to assess safety and efficacy of adoptive cell therapy with anti-PD-1 plus low-dose pegylated-interferon-alpha in patients with metastatic melanoma refractory to standard of care treatments: the ACTME trial. BMJ Open. 2020 Nov 24;10(11):e044036. doi: 10.1136/bmjopen-2020-044036. PMID 33234662